CLINICAL TRIAL: NCT06198075
Title: Effects of Action Observation Therapy on Balance in Children With Down Syndrome
Brief Title: Action Observation Therapy on Balance in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0742
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Down Syndrome
Keywords: Action Observation; Balance; Down syndrome; Rehabilitation
MeSH Terms: conditions — Down Syndrome | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study will be randomized controlled trial used to evaluate the effectiveness of action observation therapy on balance in children with down syndrome. Subjects with down syndrome meeting the inclusion and exclusion criteria will be divided into two groups using non-probability sampling technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Subjects will receive 6 weeks of general physical therapy,3 times/week for 30 min each session. The exercise program will include lying to sitting position, moving in the sitting posture, sitting and standing up, posture training for learning a normal gait pattern, weight bearing and weight movement training in the straight posture, walking training on the flat floor and stair walking. Final assessment will be done after 6 weeks
  Interventions: Other: Control Group
- Experimental group (Experimental): Subjects will watch a video on a screen from 1 meter in front of their chairs while sitting comfortably with their arms resting but they were not allowed to physically follow the video or move. The model of the video motion observation exercises will perform by the therapist and the training video consist of 4 stages that varied by difficulty and the video of each step was watched for the entire week. The participants watched a video of a task presented by the therapist and after completing the assignment they will perform the steps if step will too difficult to perform retraining will be conducted. Final assessment will be done after 6 weeks.
  Interventions: Device: Experimental Group

INTERVENTIONS:
Other: Control Group — Subjects will receive 6 weeks of general physical therapy,3 times/week for 30 min each session. The exercise program will include lying to sitting position, moving in the sitting posture, sitting and standing up, posture training for learning a normal gait pattern, weight bearing and weight movement training in the straight posture, walking training on the flat floor and stair walking. Final assessment will be done after 6 weeks
  Arms: Control group
Device: Experimental Group — Subjects will watch a video on a screen from 1 meter in front of their chairs while sitting comfortably with their arms resting but they were not allowed to physically follow the video or move. The model of the video motion observation exercises will perform by the therapist and the training video consist of 4 stages that varied by difficulty and the video of each step was watched for the entire week. The participants watched a video of a task presented by the therapist and after completing the assignment they will perform the steps if step will too difficult to perform retraining will be conducted.
  Arms: Experimental group

SUMMARY:
Down syndrome is a condition in which a child is born with an extra copy of their 21st chromosome hence its other name is trisomy 21. The hallmarks of Down syndrome are mental retardation, hypotonia and characteristic phenotype features. Balance is one of the major issue. Action observation therapy focus on the concept of balance improvement.

DETAILED DESCRIPTION:
The study will be randomized controlled trail used to evaluate the effectiveness of Action observation therapy on balance in children with down syndrome. subjects with down syndrome meeting the inclusion exclusion criteria will be divided into two groups using non-probability sampling technique. Assessment will be done using Pediatric balance scale(PBS) and Timed up and go test(TUG) . Control group will receive regular physical therapy with balance training and experimental group will receive regular physical therapy + Action observation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children with age group of 6-12
* Both male and female
* Body Mass Index (BMI) within normal range (57.1%)
* Absence of any psychiatric and physical illness at the time of participation

Exclusion Criteria:

* Uncontrolled seizures
* Any kind of orthopedic condition
* Registered visually impaired
* Severe Atlanto Axial instability
* Unable or unwilling to understand and attempt the task

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Pediatric berg balance scale | 6 weeks
  Pediatric balance scale is a modified version of berg balance scale that is used to assess functional balance skills in children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points It has good reliability and validity with (ICC=0.997) (r=0.797, p <0.05).
Modified Timed up and go test | 6 weeks
  The timed UP & GO (TUG) test was developed by Podsiadlo and Richardson in 1991 that is used to assess dynamic balance during the performance of a task. This test measures in second the time required for an individual to stand up from a standard chair with armrest, walk 3m and turn around with reliability and validity of (ICC=0.98; p<0.01).

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Jabir, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeong YA, Lee BH. Effect of Action Observation Training on Spasticity, Gross Motor Function, and Balance in Children with Diplegia Cerebral Palsy. Children (Basel). 2020 Jun 18;7(6):64. doi: 10.3390/children7060064. PMID 32570855